CLINICAL TRIAL: NCT02418910
Title: Comparative Effectiveness of Two Self Assessment Tools: KIOS-Bipolar or eMoods: A Randomized, Open 52 Week Study for Persons With Bipolar Disorder
Brief Title: Effectiveness of Two Self Assessment Tools: KIOS-Bipolar or eMoods
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Biomedical Development Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: HSC20150321
Record Dates: First submitted 2015-04-13; First posted 2015-04-17 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-08

CONDITIONS: Bipolar Disorder
Keywords: bipolar; self assessment; prospective randomized trial
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bipolar outpatients: Patients with Bipolar Disorder in any clinical state

SUMMARY:
The goal of this project is to complete the development of a patient-centered software system and mobile app to assist in managing bipolar disorder. In Phase I, the investigators developed a novel computational tool known as KIOS. Based on concepts from nonlinear systems (chaos) theory, KIOS tracks multiple interacting symptoms to determine the precise state of a BD patient. Once the patient's state is identified and the trajectory of the patient is established, KIOS produces advice specific to the patient's condition to help manage the course of the disease. To demonstrate the usability of the software, KIOS was converted to an online tool with mobile access. Twenty bipolar patients evaluated KIOS in a twelve week field trial. No technical problems with the software were observed and results showed that patients had significantly more reductions in symptom severity than increases. The development of this innovative tool to help patients self- manage BD has the potential to have a profound impact on public health and achieve significant commercial success.

DETAILED DESCRIPTION:
This Phase II study has the specific aim of evaluation of KIOS-Bipolar in a randomized, open 52 week effectiveness study of 120 bipolar subjects in current treatment at three socioeconomically diverse academic health science centers. Concurrent with this clinical effectiveness study, the research team, funded by the same NIH grant,will refine prototype software and integrate data security and establish quality standards into the KIOS-Bipolar system.

The clinical trial will:

Assess sensitivity of K-B assessed improvement or worsening by comparison with assessment by BISS-Self and BISS-42.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 18 years of age or older
2. Bipolar I or II disorder as assessed by MINI 6.0
3. In psychiatric outpatient treatment at UTHSCSA, University of Louisville, or Lindner Center of Hope, Mason Ohio
4. Currently taking mood stabilizer or second generation antipsychotic for 4 weeks or longer
5. Ability to access Kios-Bipolar or eMoods (via computer, smartphone or tablet)

Exclusion Criteria:

1. Unwilling or unable to comply with study requirements
2. Renal impairment (serum creatinine >1.5 mg/dl
3. If on thyroid medication must be euthyroid for at least 1 month
4. Drug/alcohol dependence within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This Phase II study has the specific aim of evaluation of KIOS-Bipolar in a randomized, open 52 week effectiveness study of 50 bipolar subjects in current treatment. Subjects are male or female, outpatient, 18 years of age or older, Bipolar I or II disorder as assessed by MINI 6.0, and in psychiatric outpatient treatment at UTHSCSA
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bowden, M.D., Principal Investigator — University of Texas
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bipolar Outpatients in Any Clinical State: Patients with Bipolar Disorder. Study does not provide a treatment intervention.
Period: Overall Study
Arm/Group | Bipolar Outpatients in Any Clinical State
Started | 50
Completed | 43
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Bipolar Outpatients in Any Clinical State - KIOS or eMoods: Patients with Bipolar Disorder. Study does not provide a treatment intervention.
Arm/Group | Bipolar Outpatients in Any Clinical State - KIOS or eMoods
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 43 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 33
  More than one race | 4
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Two Brief Assessment Measures: KIOS Bipolar or eMOODs
Description: measure is the count of participants with KIOS or eMOOD assessments completed on time, completed only with follow-up prompts, and the number of weeks not submitted.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bipolar Outpatients in Any Clinical State
Number analyzed (Participants) | 43
Participants | 43

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bipolar Outpatients in Any Clinical State
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02418910/Prot_SAP_000.pdf